CLINICAL TRIAL: NCT00632632
Title: Combined Exposure Therapy and D-Cycloserine vs. Placebo for Posttraumatic Stress Disorder
Brief Title: Virtual Reality & D-cycloserine (DCS) for Posttraumatic Stress Disorder (PTSD)
Acronym: VR-DCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0411007625; NCT00161499 (obsolete NCT alias)
Record Dates: First submitted 2008-02-29; First posted 2008-03-11 (Estimated); Results first posted 2015-08-27 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-07

CONDITIONS: Posttraumatic Stress Disorder
Keywords: World Trade Center Victims; Iraq War Veterans; PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Cycloserine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- D-Cycloserine (DCS) (Experimental)
  Interventions: Drug: D-Cycloserine
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: D-Cycloserine — Cognitive behavioral treatment (CBT) including prolonged exposure enhanced by virtual reality with D-Cycloserine -100 mg on days when receiving exposure with virtual reality (approximately 10-12 times)
  Arms: D-Cycloserine (DCS)
Other: Placebo — Cognitive behavioral treatment (CBT) including prolonged exposure enhanced by virtual reality. Placebo given on days when receiving exposure with virtual reality (approximately 10-12 times).
  Arms: Placebo

SUMMARY:
This study proposes to evaluate the effects of D-cycloserine (DCS) combined with Virtual Reality exposure therapy in a sample of patients who developed posttraumatic stress disorder (PTSD) following either the events of September 11, 2001, or military service in the war in Iraq. In addition, this study hopes to determine whether a common human genetic single nucleotide polymorphism (SNP) in a growth factor, brain derived neurotrophic factor, BDNF (Val66Met), predicts treatment response to PTSD.

Overall, this study aims 1) to determine if subjects administered DCS show a significantly larger decrease in symptoms of PTSD as compared to those administered a placebo, 2) to determine if subjects administered DCS show a decrease in PTSD symptomatology significantly earlier (as measured by weeks) than those administered a placebo, 3) to determine if differences in symptomatology are evident at a 6-month follow-up and indicate long-term differences between groups, and 4) to determine if the BDNF SNP predicts treatment response.

DETAILED DESCRIPTION:
Participants with 9/11-related or military service in the Iraq War-related PTSD are assigned to one of two programs, following an initial assessment. Both programs include Virtual Reality Exposure Therapy (VRET) for the treatment of PTSD as well as widely-used standard cognitive-behavioral therapy techniques. The VRET is comprised of ten ninety minute sessions which involve mental imagery as well as virtual reality presentations delivered by a special display worn over the head and eyes. The virtual reality simulations consist of either images of the World Trade Center and the events of September 11, 2001 or multiple scenarios common to military personnel assigned to Iraq. One group of participants will receive the medication cycloserine (seromycin) and one group will receive a placebo drug (like a sugar pill). Participants take a dose of medication only on the days that they come to the laboratory for the Virtual Reality Exposure (VRE) sessions, and 90 minutes prior to the VRE sessions. Some subjects in the study will receive a 100 mg dose of cycloserine, and other subjects in the study will receive the placebo (sugar pill). This will be determined randomly (as by the flip of a coin). Neither the patient nor the treating clinicians will know which pill that patients are receiving; however, this arrangement may be changed if medically necessary. Patients are briefly assessed for well-being at every session, and are reassessed following session three, session six, and session ten for changes in symptomatology. At the completion of treatment and again six months later, the principal investigator or one of her associates will reinterview participants and have them complete some questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. English-speaking adults
2. Between the ages of 18 and 70
3. Exposed to the WTC Attacks (were in towers or in the immediate area) or veterans of the Iraq War
4. Diagnosed with PTSD symptoms.

Exclusion Criteria:

1. Presence of current organic mental disorder
2. Schizophrenia
3. Bipolar disorder
4. Depression with psychotic features
5. Current substance dependence
6. Delusional disorder
7. Active suicidal ideation, intent, or plan
8. Active homicidal ideation, intent, or plan
9. Use of pacemaker
10. Medically unstable
11. Pregnant or lactating
12. A history of severe renal disease
13. History of seizures
14. Currently taking anticoagulants, ethionamide (Trecator-SC) or isoniazid (INH)
15. History of allergic reaction to cycloserine.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2005-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: JoAnn Difede, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

REFERENCES:
- See also: Related Info — http://www.patss.com

RESULTS

PARTICIPANT FLOW:
Groups:
- D-Cycloserine (DCS): D-Cycloserine: CBT including prolonged exposure enhanced by virtual reality D-Cycloserine -100 mg on days when receiving exposure with virtual reality (approximately 10-12 times)
- Placebo: placebo: Cognitive behavioral treatment including prolonged exposure enhanced by virtual reality. Placebo given on days when receiving exposure with virtual reality (10-12 times).
Period: Overall Study
Arm/Group | D-Cycloserine (DCS) | Placebo
Started | 13 | 12
Completed | 13 | 9
Not Completed | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | D-Cycloserine (DCS) | Placebo | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.77 (11.92) | 43.75 (8.72) | 45.84 (10.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 8 | 11 | 19
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 10 | 11 | 21
  Black | 1 | 0 | 1
  Hispanic | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 13 | 12 | 25

OUTCOME MEASURES:

1. Primary Outcome: Clinician Administered PTSD Scale(CAPS)
Description: Total CAPS severity score range is 0-136. Higher values represent a worse outcome (i.e. greater severity of posttraumatic symptoms). CAPS consists of 3 subscales, which are combined to form a total severity score.
  Subscales:
  CAPS cluster B (reexperiencing symptoms, range 0-40) CAPS cluster C (avoidance and numbing symptoms, range 0-56) CAPS cluster D (hyperarousal symptoms, range 0-40)
Time Frame: Immediately following treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-Cycloserine (DCS) | Placebo
Number analyzed (Participants) | 13 | 12
units on a scale | 32.38 (28.55) | 42.17 (20.75)

2. Secondary Outcome: Structured Clinical Interview for DSM-IV - Major Depressive Disorder (SCID-MDD)
Description: Structured Clinical Interview for DSM-IV - Major Depressive Disorder is a clinical interview to assess presence/absence of Major Depressive Disorder.
Time Frame: Immediately following treatment
Measure: Number; unit: percentage of MDD remission
Arm/Group | D-Cycloserine (DCS) | Placebo
Number analyzed (Participants) | 13 | 12
percentage of MDD remission | 78 | 60

3. Primary Outcome: Clinician Administered PTSD Scale(CAPS)
Description: as for outcome 1
Time Frame: 6-months follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-Cycloserine (DCS) | Placebo
Number analyzed (Participants) | 13 | 12
units on a scale | 24.15 (26.48) | 45.92 (25.66)

ADVERSE EVENTS:
Arm/Group | D-Cycloserine (DCS) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 0/13 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes